CLINICAL TRIAL: NCT04495361
Title: A Pedagogical Research on Use of an Online Learning Platform by Final Year Medical on Under Five Pneumonia
Brief Title: Online Learning Portal on Under Five Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Maternal, Neonatal and Child Health Research Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16/136/108
Record Dates: First submitted 2020-04-17; First posted 2020-07-31 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Pneumonia; Childhood Pneumonia; Infectious Disease; Acute Respiratory Infection
Keywords: Childhood Pneumonia; Acute respiratory illness; Pakistan
MeSH Terms: conditions — Pneumonia; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Students will be exposed to an online learning portal in which they will undergo planned electronic encounters with under five patients having pneumonia. For each case, students will have to identify the category of pneumonia and the appropriate treatment/ management in a timed session.
  Upon clicking on the available case, the participant will be shown a typical case of either no pneumonia, pneumonia or severe pneumonia. The video will run for around thirty seconds to one minute during and after which the students will try to identify the case and select its category from the drop down menu of diagnosis. There will be tabs for history, examination, diagnosis and management. The student will select the best suited response from a range of options. Based on the selection of the response and the time taken to do so, a score will be generated. The student can take two attempts for each case. Students will be required to a login for 6 months whereby 3 cases will be assigned per month.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online learning portal (Experimental): Final year medical students will use an online learning portal in which three case scenarios of under five pneumonia patients will be displayed each month. Based on history and examination, the user will diagnose and manage the patient.
  Interventions: Other: E-learning portal

INTERVENTIONS:
Other: E-learning portal — An online learning portal for the identification and management of pneumonia in under five children

SUMMARY:
Despite the availability of standard pneumonia management guidelines and multiple global efforts, pneumonia continues to be the leading killer of children under five, accounting to around 17% of the total under five deaths globally. In Pakistan, pneumonia contributes to 16% of under five mortality in the country having a well-defined yet poorly functional healthcare system.

Although, there are standard set of guidelines for management of pneumonia patients however, the management practices of this illness are variable across the country. This could be attributed to non-availability of work ready graduates which in turn is due to variations of teaching methods across various institutions. Although the medical students across these institutions do get exposed to clinical cases in the final year however, this exposure is also variable. If this clinical experience is coupled with an adjunct capacity building mode using an online platform. there is a possibility that students could be trained in a better way.

DETAILED DESCRIPTION:
The investigators plan to use e-learning portal in identification and management of under five pneumonia cases as it is one of the leading killers of children under five which is largely managed non-uniformly across the country. The investigators will use videos of patients under five years of age with pneumonia and allow virtual performance of clinical skills by medical students in an online platform. Such a platform can prove to be an adjunct to standard clinical education rather than a substitute. The investigators propose that this platform will help the medical students to prepare them for a range of clinical challenges as it is an ideal strategy for the development, refinement, and rehearsal of skills in recognition in a safe environment.

Primary Objective: To measure final year medical student's theoretical (knowledge) and applied (virtual clinical performance) learning on under five pneumonia case management in an e-learning package

Secondary Objective: To explore associations between student characteristics and outcomes following exposure to the e-learning program

Study design: This will be a multi-center quasi experimental study with final year medical students studying in various institutions in the twin cities of Pakistan (Islamabad/Rawalpindi).

The design of the package will be based on the FIRST2ACT Web platform which is an e-learning platform for medical students which focuses on exposure of the users to different adult simulated case scenarios in the form of videos.

Three categories of case scenarios, based on WHO classification of pneumonia, will be presented to the students. Thus case scenarios of patients with no pneumonia, pneumonia and severe pneumonia will be presented.

Stages of study: The study will be conducted in the following three stages all of which will be mostly conducted electronically.

Pre-intervention stage:

Piloting of existing resources: The case scenarios will be created of children under five suffering from pneumonia. The host organization MNCHRN has an archive of different videos of patients of pneumonia already available which have been developed as a part of another activity. Consent forms from the caregivers of the patients in the videos including permission to use them in future for other purposes are in the record. These videos after testing will be incorporated in the program. If it is felt that the existing content does not fulfil the purpose, then new videos will be recorded of under five pneumonia cases in a hospital facility by taking consent from the caregivers.

Development of new cases: If required, new videos showing different types of pneumonia in under five children visiting a clinic or admitted in a hospital will be recorded. Approval from the clinic/ hospital will be taken to include their patients and to record videos in their premises. Consent from the carers/parents to videotape their children would also be taken. Details on the purpose of the study and their participation will be explained to them and will also be provided in written form prior to signing the consent form.

Development and testing of portal: Who, how, where, what framework shall be employed for the development and implementation of the e-learning package. An expert of IT will be recruited for the development of portal. Portal will be tested by the research team, medical students and paediatricians.

Invitation to institutions to participate: The heads of each institution will be approached to provide permission for involvement of their final year medical students. Approval and ethical clearance from institution's research committees will be taken.

Introductory seminar: After approval, seminars for final year medical students to facilitate their participation in the study will be conducted in each institution. Purpose of the study and the use of portal will be explained to them. Information sheets and consent forms will be distributed to the students at the end of the seminar and they will be given one week to consider the information and decide if they want to participate.

Participant's consent and enrolment: Name of the student and institution, age, gender, phone number, email address will be taken from the interested students at the time of enrolment in the study. Once enrolled, the students will be informed that a login ID to access the e learning platform will be provided at their email addresses. The same login ID will be used as the participant's identifier and the means of linking individual data throughout the study.

The following online questionnaires will be filled in by the enrolled students after they log on to the portal for the first time.

1. Demographic and clinical experience
2. Pre-test self-assessment of knowledge, skills, confidence, and competence

Study debriefing: Each participant will be able to access a narrated PowerPoint presentation on the intervention with instructions within the portal. The briefing will describe the approach and scenarios in general with examples the participants would see and instructions on selecting clinical actions and receiving feedback. It will also explain the parameters (number of attempts and time taken to complete the case scenario) that will be accounted in the scoring.

Intervention stage:

Exposure on online clinical cases: This will be an online program; therefore the students will be able to access it anywhere and anytime they feel convenient provided there is internet connectivity. In case there is interruption of internet due to electricity shortage, efforts will be made to keep the interface such that the students takes up from where they left provided the shortage is not of more than one hour as the student might forget some components of the training.

Students after log in to the portal will undergo a planned electronic encounter with an under five patient suffering from pneumonia. For each case, students will have to identify the category of pneumonia and the appropriate treatment/ management in a timed session The interface will be developed such that upon login, the student will be given an opportunity to select cases. Upon clicking on the icon of the age group, the participant will have a screen popping up showing a typical case of either no pneumonia, pneumonia or severe pneumonia. The video will run for around thirty seconds to one minute during and after which the students will try to identify the case and select it from the drop down menu of whether it is no pneumonia, pneumonia or severe pneumonia. There will be tabs for history, examination, diagnosis and management. The student will select the best suited response from a range of options.Based on the selection of the response and the time taken to do so, a score will be generated. The student can take three attempts for each case scenario. The total score will be an average of all attempts.

Feedback on the scored performance: Based on the score the student will be provided with general formative feedback incorporating patient diagnosis and best practice management for that case.

The intervention will continue for six months with instructions to log in every month.

Post-intervention stage: Participants will complete the knowledge post-test and a self-evaluation of skills, competence and confidence in managing under five patients after the intervention. The overall performance of each student will be scored and students will receive a summarized feedback and provided with links to resources for further self-directed learning. Finally, they will complete an evaluation of their experience and receive a printable certificate of completion.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for medical students:

* Final year medical students studying in institutions in Rawalpindi/Islamabad registered under the higher education commission
* Medical students whose heads have provided permission to undertake the study with them
* Medical students who have provided a written consent to be included in the study.

Inclusion Criteria for pneumonia patients

* Patients less than five years diagnosed with no pneumonia, pneumonia or severe pneumonia
* Parents/Carers who provide consent for their under five children to be videotaped.

Exclusion Criteria:

Exclusion Criteria fro medical students

* Medical students withdrawing/leaving the institute
* Medical students who are not in final year

Exclusion Criteria for pneumonia patients

* Patients under five suffering from comorbidity with pneumonia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline knowledge of all participants on under five pneumonia at 6 months | 6 months
  Self administered questionnaire with multiple choice questions will be filled by the participants. 1 score for each correct response and 0 for incorrect response will be given.
Change from baseline confidence in skills of all participants in diagnosing and managing under five pneumonia at 6 months | 6 months
  Self-administered Likert scale questionnaire where 1 means low and 5 high will be filled by the participants

CONTACTS AND LOCATIONS:
Overall Officials: Dr Tabish Hazir, MBBS, FRCPCH, Principal Investigator — Maternal, Neonatal and Child Health Research Network
Locations (1):
- MNCHRN, Islamabad, Federal, Pakistan